CLINICAL TRIAL: NCT02491138
Title: An Evaluation of Appearance-based Interventions for the Promotion of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Collaborators: Duke-NUS College (Unknown); University of St Andrews (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-15-083
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2017-07

CONDITIONS: Sleep Habits; Healthy
Keywords: participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard information (Placebo Comparator): In this arm, participants will receive standard information pamphlets about the benefits of good sleeping habits.
  Interventions: Other: Pamphlets
- Appearance-based information (Experimental): In this arm, participants will receive information about how sleep modifies their physical appearance. This will involve a computer transformation that morphs their face according to hours of sleep obtained.
  Interventions: Behavioral: Appearance-based intervention

INTERVENTIONS:
Behavioral: Appearance-based intervention
  Arms: Appearance-based information
Other: Pamphlets
  Arms: Standard information

SUMMARY:
This study evaluates the efficacy of appearance-based interventions in promoting healthy sleep. One group of participants will receive standard information about sleep (control group), while the other group will receive information about how sleep affects their physical appearance (intervention group).

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years
* <7 hours of sleep routinely

Exclusion Criteria:

* per-existing medical, sleep, or psychiatric conditions;
* history of substance abuse.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Objective sleep duration | Up to 1 month after the intervention
  Measured through actigraphy
Self-reported sleep hygiene | Up to 1 month after the intervention
  Measured through the Sleep Hygiene scale (total score: higher score corresponds to poorer sleep hygiene)

SECONDARY OUTCOMES:
Subjective sleep quality | Up to 1 month
  Measured through the Pittsburgh Sleep Quality Index (global score: higher score corresponds to poorer sleep quality)
Insomnia-related cognition | Up to 1 month
  Measured through the Dysfunctional Beliefs and Attitudes about Sleep scale (total score: higher score corresponds to more dysfunctional beliefs and attitudes)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

REFERENCES:
- [Derived] Perucho I, Vijayakumar KM, Talamas SN, Chee MW, Perrett DI, Liu JCJ. A Web-Based Photo-Alteration Intervention to Promote Sleep: Randomized Controlled Trial. J Med Internet Res. 2019 Sep 26;21(9):e12500. doi: 10.2196/12500. PMID 31573913